CLINICAL TRIAL: NCT05389215
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of DWN12088 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of DWN12088 in Patients With IPF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWN12088201
Record Dates: First submitted 2022-04-17; First posted 2022-05-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — BID protein, human; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DWN12088 Xmg Tablet (BID) (Experimental): PRS inhibitor
  Interventions: Drug: DWN12088
- Placebo 0mg Tablet (BID) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWN12088 — DWN12088 Xmg Tablet (BID)
  Other Names: DWN12088 Xmg Tablet (BID)
  Arms: DWN12088 Xmg Tablet (BID)
Drug: Placebo — Placebo 0mg Tablet (BID)
  Other Names: Placebo 0mg Tablet (BID)
  Arms: Placebo 0mg Tablet (BID)

SUMMARY:
This is a randomized, double-blinded, placebo-controlled multicenter study to evaluate the safety and efficacy of DWN12088 in patients with Idiopathic Pulmonary Fibrosis.

DETAILED DESCRIPTION:
This is randomized, double-blinded, placebo-controlled multicenter study to evaluate the safety and efficacy of DWN12088 in patients with Idiopathic Pulmonary Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥40 years based on the date of the written informed consent form
* Diagnosis of IPF as defined by American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines
* In a stable condition and suitable for study participation based on the results of medical history, physical examination, vital signs, 12-lead ECG, and laboratory evaluation
* Patients receiving local standard-of-care for IPF, defined as either pirfenidone or nintedanib, at a stable dose for at least 3 months prior to screening, or neither pirfenidone nor nintedanib. If the patients were on pirfenidone or nintedanib previously and have been off for at least 3 months prior to screening, they will be considered as not on any treatment for IPF
* Meeting all of the following criteria during the screening period:

  * FVC ≥40% predicted of normal
  * DLCO corrected for Hgb ≥25% and ≤80% predicted of normal.
  * forced expiratory volume in the first second/FVC (FEV1/FVC) ratio ≥0.7 based on pre-bronchodilator value

Exclusion Criteria:

* Acute IPF exacerbation within 6 months prior to screening and/or during the screening period
* Patients who are unwilling to refrain from smoking within 3 months prior to screening and until the end of the study
* Female patients who are pregnant or nursing
* Abnormal ECG findings
* Use of any investigational drugs for IPF within 4 weeks prior to screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of decline of FVC | From Day 1 through Week 24
  To investigate the efficacy of DWN12088 on pulmonary function
Incidents of treatment-emergent adverse events | From Day 1 through Week 24
  To evaluate the safety and tolerability of DWN12088 compared with placebo

SECONDARY OUTCOMES:
Time to progression of IPF | From Day 1 through Week 24
  To evaluate the efficacy of DWN12088 on time to progression of IPF
Quantitative high-resolution computed tomography | From Day 1 through Week 24
  To evaluate the efficacy of DWN12088 as measured by quantitative high-resolution computed tomography
Functional exercise capacity, assessed by the 6-minute walk test (6MWT) distance | From Day 1 through Week 24
  To evaluate the efficacy of DWN12088 on functional exercise capacity, assessed by 6MWT distance
Diffusing capacity of lung for carbon monoxide (DLCO) corrected for Hgb | From Day 1 through Week 24
  To evaluate the efficacy of DWN12088 on pulmonary diffusion function

CONTACTS AND LOCATIONS:
Overall Officials: Song, Principal Investigator — AIDS Malignancy Consortium
Locations (30):
- United States (20):
  - Pulmonary Associates, PA, Mesa, Arizona
  - Dignity Health Norton Thoracic Institute, Phoenix, Arizona
  - The University of California San Francisco, San Francisco, California
  - Loyola University Medical Center (LUMC), Maywood, Illinois
  - University of Kansas Medical Center Research Institute, Inc, Kansas City, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Michigan Center, Michigan
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Pulmonix Research, LLC, Greensboro, North Carolina
  - Legacy Research Institute, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The U.S. Department of Veterans Affairs, Charleston, South Carolina
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health San Antonio Medical Arts & Research Center, San Antonio, Texas
- South Korea (10):
  - Inje University Busan Paik Hospital, Busan, Busan
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggido
  - Ajou University Hospital, Hwaseong-si, Gyeonggido
  - Seoul National University Hospital, Seoul, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Ulsan University Hospital, Ulsan, Ulsan

IPD SHARING:
Plan to Share IPD: No